CLINICAL TRIAL: NCT04011514
Title: Specialized Stroke Unit Nursing Interventions in the Emergency Department and Their Efficacy on Outcomes and Patient Perceptions of Clinical Care Pathway Coherence
Brief Title: Querying Stroke Unit Nursing Interventions in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Senior consultant and faculty supervisor, DMSc, Ph.D.,, Herlev Hospital
Other Study IDs: H-17035544
Record Dates: First submitted 2018-10-20; First posted 2019-07-08 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-01

CONDITIONS: Stroke; TIA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline period: Usual care. Stroke patients admitted to the ED during the 3-month baseline inclusion period.
  Interventions: Behavioral: Dedicated stroke nurse care in ED
- Intervention period: Intervention: 2 month implementation period of specialized stroke nurses allocated to ED for nurse specific treatment of stroke patients specific observations and care
  Interventions: Behavioral: Dedicated stroke nurse care in ED

INTERVENTIONS:
Behavioral: Dedicated stroke nurse care in ED — A specialized SU nursing team partner with ED nursing staff for timely fulfillment of stroke quality care indicators while awationg admission to a dedicated stroke unit

SUMMARY:
The aim of the study is to monitor if specialized stroke nurses as team partners in the ED can reduce hospital acquired infections. The study is designed as pre- post-intervention study in which specialized SU nurses partner with ED nursing staff to asses and screen stroke admissions in the ED.

DETAILED DESCRIPTION:
An intervention study comprised of 1) a primary registry database component and 2) a secondary questionnaire based quantitative evaluation . The intervention study includes a 3-month baseline observational period followed by a 7-month baseline data collection period, a 2-month intervention implementation phase, and a 3-month intervention observational period followed by 7-month intervention data collection period.

An intervention, where dedicated stroke nurses handle acute care of stroke and TIA patient in the ED prior to admission to a dedicated stroke unit will take place in the timeframe of 11-19:00 hrs, 7 days a week. Notably, the intervention is set to be integrated into clinical practice on a permanent basis after end of study.

Data for all stroke patients admitted to the ED at HGH are collected during the 3-month baseline and intervention observational periods. Fulfilment of Danish Stroke Quality Program (DAP) quality indicators is monitored as follows - use of dysphagia screen (GUSS), mobilization within day of ED admission and transfer to SU. Additional nursing interventions monitored in the ED are: Use of nasogastric catheter, use of bladder scan and intermittent catheterization, frequency of temperature monitoring and use of anti-pyretics, acute phase monitoring of blood-pressure every 2 hours, use of Scandinavian Stroke Scale (SSS) score.

Outcomes are monitored in hospital and at visits to the out patient clinic, as well as by registry.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the ED at Herlev Hospital with a diagnosis of stroke or TIA from 11 Am to 7 PM
* patients fulfilling one of the following ICD-10 codes at discharge: ICH: I61, cerebral infarction; I63, unspecified: I64, TIA: G45 and a scheduled follow-up appointment at the outpatient clinic Herlev Hospital

Exclusion criteria:

* Patients transferred from other hospitals or stroke units
* Patients elegible for thrombolysis or thrombectomy at time of admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted with a diagnosis of acute stroke or TIA and candidate to specific stroke observation within the following 24 hours minimum.
  Data for all stroke/TIA patients admitted to the ED at HGH are retrieved during the 3-month baseline and a 3 month intervention observational period during admission and at regular clinical follow-up.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-09-21 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections | 7 days from admission
  Incidence of pneumonia and urinary tract infections defined by a combination of clinical symptoms and para-clinical tests.

SECONDARY OUTCOMES:
30-day mortality or recurrent cerebrovascular event | 30 days from first admission
  Composite measure of mortality, cerebrovascular or cardiovascular incidence
Rate of re-admission within 30 days | 30 days from first admission
  Number of re-admission for any disease post stroke
Number of patients with post stroke depression | baseline and 90 days and 1 year after admission
  new onset depression and antidepressant prescriptions within 90 days and 1 year from stroke
Level of 90-day post-stroke dependency | baseline and 90 days from admission
  via modified Rankin Scale (mRS) score (0-6, 0=best)
Mental health | within 90 days from admission
  WHO-Five Well-Being index
Length of stay | 90 days from admission
  Total time of hospital admission
Dependency | Within 90 days from admission
  Barthel Index

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD, DMSc, Principal Investigator — Department of Neurology, Herlev-Gentofte Hospital
Locations (1):
- Department of Neurology, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participants data cannot be shared with 3rd parties as these data are protected by danish law.